CLINICAL TRIAL: NCT01239511
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Dose-Response and Safety of STA-2 in Patients With Chronic Stable Angina
Brief Title: Phase IIb Study of STA-2 in Patients With Chronic Stable Angina
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinphar Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCCD09004A
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — Tea; STA 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo group (Placebo Comparator): placebo capsule 2# t.i.d./day
  Interventions: Drug: green tea polyphenols (STA-2)
- Treatment Group A (Experimental): 150 mg STA-2, 2 capsules t.i.d., after meal (900 mg STA-2 total dose per day)
  Interventions: Drug: green tea polyphenols (STA-2)
- Treatment Group B (Experimental): 300 mg STA-2, 2 capsules t.i.d., after meal (1800 mg STA-2 total dose per day)
  Interventions: Drug: green tea polyphenols (STA-2)
- Treatment Group C (Experimental): 450 mg STA-2, 2 capsules t.i.d., after meal (2700 mg STA-2 total dose per day)
  Interventions: Drug: green tea polyphenols (STA-2)

INTERVENTIONS:
Drug: green tea polyphenols (STA-2) — 2 capsules t.i.d., after meal

SUMMARY:
The objective of this study is to evaluate the dose-response of three different dose levels of STA-2 (900 mg daily, 1800 mg daily and 2700 mg daily for 42 days) versus placebo in patients with chronic stable angina.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the dose-response of three different dose levels of STA-2 (900 mg daily, 1800 mg daily and 2700 mg daily for 42 days) versus placebo in patients with chronic stable angina.

Treatment Group A:

150 mg STA-2, 2 capsules t.i.d., after meal (900 mg STA-2 total dose per day)

Treatment Group B:

300 mg STA-2, 2 capsules t.i.d., after meal (1800 mg STA-2 total dose per day)

Treatment Group C:

450 mg STA-2, 2 capsules t.i.d., after meal (2700 mg STA-2 total dose per day)

Placebo Group:

Placebo capsule, 2 capsules t.i.d., after meal

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≧ 20 years;
2. Subjects weight > 50 kg
3. subjects who had more than 50% coronary stenosis documented by catheterization or ever received coronary intervention;
4. The two ETT results at screening (Visit 1) and baseline (Visit 2) show greater than or equal to 1 mm ST-segment depression within exercise duration;
5. The difference in exercise duration between screening (Visit 1) and baseline (Visit 2) do not exceed 20% of the longer test;
6. Able to provide written informed consent.

Exclusion Criteria:

1. Subjects with pacemaker rhythm, unstable angina or myocardial infarction within the preceding 3 months;
2. Subjects with heart failure (New York Heart Association class III or IV), uncorrected valvular or congenital heart disease, subjects who need digoxin or digitalis;
3. Subjects with any resting EKG abnormalities preventing the interpretation of ischemia as judged by the investigator;
4. Subjects with COPD requiring bronchodilators;
5. Subjects with impaired hepatic function (defined as AST or ALT > 2X the upper limit of normal values), or impaired renal function (defined as serum creatinine > 1.5 mg/dL), or diagnosis of any chronic renal/hepatic disease;
6. Subjects with documented evidence of gastroduodenal ulcer disease, gastrointestinal bleeding or other gastrointestinal disease within the preceding 3 months as judged by investigator;
7. Subjects who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with safety assessments during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, immune, neurological, or hematological disease as determined by the clinical judgment of the investigator;
8. Subject with any conditions that could interfere the performance of exercise tolerance test as judged by investigator (e.g., knee/ankle arthropathy, Parkinsonism, stoke);
9. Female subjects of childbearing potential who:

   * are lactating;
   * have positive pregnancy test (urine) at V1;
10. Subject has received any investigational agent within 28 days prior to the first dose of investigational product;
11. Subjects who have had administered STA-2 in prior clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Den Tseng, MD, Ph.D, Principal Investigator — Department of Cardiology National Taiwan University Hospital
Locations (5):
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan
  - Chi Mei Medical Center, Tainan, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - Taipei Medical University-Shuang Ho Hospital, Taipei, Taiwan
  - Taipei Veterans General Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from Nov. 2010 through Apr. 2012. There are 5 study sites participated in this study, including National Taiwan University Hospita, Chi Mei Medical Center, Taipei Veterans General Hospital, Taipei Medical University-Shuang Ho Hospital and Kaohsiung Medical University Chung-Ho emorial Hospital.
Pre-assignment Details: In order to ensure the consistency, the difference of total exercise time between V1 and V2 should be less than 20%.
Period: Overall Study
Arm/Group | Placebo Group | Treatment Group A | Treatment Group B | Treatment Group C
Started | 47 | 45 | 47 | 47
Completed | 46 | 40 | 43 | 38
Not Completed | 1 | 5 | 4 | 9

BASELINE CHARACTERISTICS:
Population: For subjects without the primary efficacy variable due to early discontinuaton and those with protocol violation were excluded from the analysis group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Treatment Group A | Treatment Group B | Treatment Group C | Total
Number analyzed (Participants) | 46 | 43 | 42 | 37 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 24 | 30 | 23 | 106
  >=65 years | 17 | 19 | 12 | 14 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (0.76) | 62.1 (10.40) | 61.4 (10.57) | 59.6 (10.11) | 61.0 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 4 | 28
  Male | 37 | 36 | 34 | 33 | 140
Region of Enrollment [Number; unit: participants]
  Taiwan | 46 | 43 | 42 | 37 | 168

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Exercise Time (Seconds)
Description: the time difference of total exercise time from V2 to V5 compare to placebo
Time Frame: 6 weeks after the first exercise tolerance testing is conducted
Population: ITT (intend-to-treat) population will be used for analysis
Measure: Least Squares Mean (Standard Deviation); unit: second
Arm/Group | Placebo Group | Treatment Group A | Treatment Group B | Treatment Group C
Number analyzed (Participants) | 46 | 43 | 42 | 37
second | 24.3 (8.73) | 18.2 (8.95) | 33.9 (9.03) | 11.9 (9.69)

2. Secondary Outcome: Change in Time to Onset of Angina From Baseline to the Final Visit
Time Frame: 6 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Time to 1mm ST-segment Depression During ETT From Baseline to Final Visit
Time Frame: 6 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Time to Maximum ST-segment Depression During ETT From Baseline to the Final Visit
Time Frame: 6 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Changes in Angina Frequency in Subject's Diary From Baseline to All Visits
Time Frame: 6 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change in Consumption of Short-acting Nitrates From Baseline to All Visits
Time Frame: 6 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change in Pharmacological Parameters (Oxidized-LDL), Isoprostane and High-sensitivity Hs-CRP From Baseline to All Visits
Time Frame: 6 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Change in Lipid Profiles (HDL-C, LDL-C, Total Cholesterol, Triglyceride) From Baseline to All Visits
Time Frame: 6 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Dose-response Relationship of Three Different Dose Levels of STA-2 Versus Placebo Control in Change in Total Exercise Time.
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo Group | Treatment Group A | Treatment Group B | Treatment Group C
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/45 | 2/47 | 1/47
Other Adverse Events (participants affected / at risk) | 0/47 | 2/45 | 2/47 | 1/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=47) | Treatment Group A (N=45) | Treatment Group B (N=47) | Treatment Group C (N=47)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Group (N=47) | Treatment Group A (N=45) | Treatment Group B (N=47) | Treatment Group C (N=47)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No